CLINICAL TRIAL: NCT04619134
Title: Effects of Non Pain Contingent Spine Rehabilitation Therapy in Chronic Low Back Pain
Brief Title: Non Pain Contingent Spine Rehabilitation Therapy in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00673 Fariha Altaf
Record Dates: First submitted 2020-11-01; First posted 2020-11-06 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Non Pain Contingent Spine Rehabilitation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NCSR Program (Experimental): Non Pain Contingent Spinal Rehabilitation
  Interventions: Other: NCSR Program
- Conventional Physical therapy (Active Comparator): Conventional Physical Therapy
  Interventions: Other: conventional physical therapy

INTERVENTIONS:
Other: NCSR Program — flexibility exercise,strengthening exercise,dynamic strengthening exercise,endurance training,counselling session
  Arms: NCSR Program
Other: conventional physical therapy — hot pack,flexibility training,strengthening exercise.
  Arms: Conventional Physical therapy

SUMMARY:
The aim of study is to determine effects of non pain contingent spine rehabilitation in chronic low back pain.A Randomized controlled trial will be conducted at Railway general hospital.

Sample size will be 32.Participants will be divided in two groups, 16 participants in group A will receive Non pain contingent spine rehabilitation (NCSR) therapy and 16 Group B will receive conventional physical therapy. The study duration will be six months. Purposive non probability sampling technique will be applied.

DETAILED DESCRIPTION:
Low back pain is defined as pain and discomfort below the costal margin and above the inferior gluteal folds. It has different characteristics such as aching, burning, stabbing, sharp or dull, well-defined, or vague. Low back pain may have intensity varying from mild to severe . Low back pain (LBP) causes more disability than any other medical condition worldwide Low Back Pain has a significant impact on functional capacity, as pain restricts occupational activities and is a major cause of absenteeism. Chronic low Back pain is defined as chronic when pain remains for more than three months it has different characteristics. Many authors define chronic pain as pain that lasts beyond the expected period of healing. Low back pain is classified and treated according to duration of symptoms, cause, absence or presence of radiculopathy and associated anatomical and radiographic changes. Symptoms persisting for less than 4 weeks is defined as acute low back pain and in sub-acute low back pain symptoms lasts for 4-12 weeks, chronic low back pain lasts for more than 12 weeks. Back pain can also be categorized into specific and nonspecific back pain, Specific back pain has a specific cause for example fracture and infection etc. and nonspecific is of unknown etiology. Non-specific pain is most common type of back pain. The prevalence of low back pain has been reported among many people especially when resulting from work related and occupational activities 75-84% of the general population suffer from low back pain and among them, it is estimated that 5-10% of the people experience LBP resulting in severe morbidity, increased health care costs, sick leaves and individual suffering. Men and women are equally reported to be affected by this condition. Core muscles maintain spinal stability, first group include deep core muscles also called local stabilizing muscles primarily include the transversus abdominis, lumbar multifidus, internal oblique muscle and quadratus lumborum. Second group include shallow core muscles, also known as global stabilizing muscles, including the rectus abdominis, internal and external oblique muscles, erector spinae, quadratus lumborum, and hip muscles. The causes of chronic low back pain are complex, several of which are unknown one major cause involves the weakening of the shallow trunk and abdominal muscle, another cause of chronic low back pain is the weakening of deep trunk muscles, such as the lumbar multifidus and transversus abdominis. Patients usually experience pain during lifting it leads to avoidance behavior and cause disability. Less intensive and cost effective non pain contingent rehabilitation therapy could target fear avoidance behavior toward lifting and in restoration of normal function.

In female patients with chronic low back pain, Primary outcome measures were recorded by visual analogue scale (VAS) and oswestry disability index (ODI) .Patterns of improvement suggested that the Non pain Contingent Spinal Rehabilitation approach is more effective than Conventional Physical Therapy in female patients with chronic low back pain. It is feasible to adapt progressive Isoinertial lifting evaluation for determining the lifting capacity, it is a valid and reliable method. Lumbar dynamic strengthening exercises are beneficial in the treatment of chronic nonspecific LBP for reduction of pain, improvement in functional ability, increase range of motion and improve core strength. Exercise intervention programs involving either muscular strength, flexibility or aerobic fitness is beneficial for nonspecific chronic low back pain. Effects of lumbar stabilization exercise on functional disability and lumbar lordosis angle in patients with chronic low back pain in 2015 Lumbar stabilization exercise and conservative program were performed 3 times a week for 6 weeks and he reported that lumbar stabilization exercise is more effective than conservative treatment for improving functional disability and lumbar lordosis angle, and significant decrease in Oswestry disability index score. Comparative effect of core muscles strength training with supine bridging over prone bridging in patients with nonspecific low back pain and concluded that prone bridging exercise is more effective in improvement of functional activities and reducing pain than supine bridging exercise program in nonspecific low back pain. Effectiveness of core stabilization exercises and routine exercise therapy in management of pain in chronic non-specific low back pain" in which he reported that Core stabilization exercise is more effective than routine physical therapy exercise in terms of greater reduction in pain in patients with non-specific low back pain. In 2013 The purpose of the study was to determine the effect of core stabilization exercises in comparison with conventional exercises on pain, functional status in patients with non-specific LBP and they concluded Core stabilization exercises found to be more effective in reducing pain and improving functional status by decreasing disability of patients with non-specific low back pain in comparison with conventional exercises. Progressive Isoinertial Lift Evaluation (PILE) method was developed by Mayer et al.in PILE protocol describes it as lifting of weight in a box from floor to waist (lumbar test) or from floor to shoulder height (cervical test) at a rate of four lifts in a 20 second interval.

ELIGIBILITY:
Inclusion Criteria:

* Patient with non-specific chronic low back pain(>3months)

Exclusion Criteria:

* Spinal surgery
* Compression Fracture
* Disc Herniation
* Cauda equina
* Pregnancy
* Cancer
* Progressive neurological disorder
* Any Psychological disorder

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 6th week
  Visual analogue scale (VAS) is a simple and frequently used method for the assessment of variations in intensity of pain. The VAS consists of a 10cm horizontal line with the words "no pain" and "worst pain" at the line's end. VAS is a reliable and valid tool to reliable and valid tool to measure pain intensity measure pain intensity. Changes from the baseline will be measured and at 4th week and then at 6th week
Functional Disability: Oswestry Disability Index | 6th week
  The Oswestry Disability Index (ODI) is one of the most commonly used outcome measures for the evaluation and treatment of LBP and it is valid, reliable. Changes from the baseline will be measured and at 4th week and then at 6th week

SECONDARY OUTCOMES:
Lumbar Range of Motion | 6th week
  Bubble Inclinometer. Changes from the baseline will be measured and at 4th week and then at 6th week
Shirado test: to assess isometric endurance of trunk flexors | 6th week
  To evaluate "flexor endurance" Patient in supine position asked to raise the lower extremities with 90 degrees flexion at hip and knee joint and also maintain cervical flexion, maintain this position for at least 5 minutes. Changes from the baseline will be measured and at 4th week and then at 6th week
Ito test: to evaluate isometric endurance of trunk extensors | 6th week
  To measure "extensor endurance" patient in prone position holding sternum off the treatment table and a small pillow below abdomen to decrease lordosis; and maintaining cervical flexion with pelvic stabilization and gluteal contraction maintain this position for 5 minutes. Changes from the baseline will be measured and at 4th week and then at 6th week
Lifting endurance | 6th week
  Progressive Iso inertial lifting evaluation(PILE). Changes from the baseline will be measured and at 4th week and then at 6th week
Fear Avoidance Belief Questionnaire | 6th week
  Fear Avoidance Belief Questionnaire (FABQ). Changes from the baseline will be measured and at 4th week and then at 6th week

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gordon R, Bloxham S. A Systematic Review of the Effects of Exercise and Physical Activity on Non-Specific Chronic Low Back Pain. Healthcare (Basel). 2016 Apr 25;4(2):22. doi: 10.3390/healthcare4020022. PMID 27417610
- [Background] Qaseem A, Wilt TJ, McLean RM, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Denberg TD, Barry MJ, Boyd C, Chow RD, Fitterman N, Harris RP, Humphrey LL, Vijan S. Noninvasive Treatments for Acute, Subacute, and Chronic Low Back Pain: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2017 Apr 4;166(7):514-530. doi: 10.7326/M16-2367. Epub 2017 Feb 14. PMID 28192789
- [Background] Nijs J, Apeldoorn A, Hallegraeff H, Clark J, Smeets R, Malfliet A, Girbes EL, De Kooning M, Ickmans K. Low back pain: guidelines for the clinical classification of predominant neuropathic, nociceptive, or central sensitization pain. Pain Physician. 2015 May-Jun;18(3):E333-46. PMID 26000680
- [Background] Chang WD, Lin HY, Lai PT. Core strength training for patients with chronic low back pain. J Phys Ther Sci. 2015 Mar;27(3):619-22. doi: 10.1589/jpts.27.619. Epub 2015 Mar 31. PMID 25931693
- [Background] Bhadauria EA, Gurudut P. Comparative effectiveness of lumbar stabilization, dynamic strengthening, and Pilates on chronic low back pain: randomized clinical trial. J Exerc Rehabil. 2017 Aug 29;13(4):477-485. doi: 10.12965/jer.1734972.486. eCollection 2017 Aug. PMID 29114516
- [Background] Cho I, Jeon C, Lee S, Lee D, Hwangbo G. Effects of lumbar stabilization exercise on functional disability and lumbar lordosis angle in patients with chronic low back pain. J Phys Ther Sci. 2015 Jun;27(6):1983-5. doi: 10.1589/jpts.27.1983. Epub 2015 Jun 30. PMID 26180363
- [Background] Akhtar MW, Karimi H, Gilani SA. Effectiveness of core stabilization exercises and routine exercise therapy in management of pain in chronic non-specific low back pain: A randomized controlled clinical trial. Pak J Med Sci. 2017 Jul-Aug;33(4):1002-1006. doi: 10.12669/pjms.334.12664. PMID 29067082
- [Background] Inani SB, Selkar SP. Effect of core stabilization exercises versus conventional exercises on pain and functional status in patients with non-specific low back pain: a randomized clinical trial. J Back Musculoskelet Rehabil. 2013;26(1):37-43. doi: 10.3233/BMR-2012-0348. PMID 23411647
- [Background] Ito T, Shirado O, Suzuki H, Takahashi M, Kaneda K, Strax TE. Lumbar trunk muscle endurance testing: an inexpensive alternative to a machine for evaluation. Arch Phys Med Rehabil. 1996 Jan;77(1):75-9. doi: 10.1016/s0003-9993(96)90224-5. PMID 8554479
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Saur PM, Ensink FB, Frese K, Seeger D, Hildebrandt J. Lumbar range of motion: reliability and validity of the inclinometer technique in the clinical measurement of trunk flexibility. Spine (Phila Pa 1976). 1996 Jun 1;21(11):1332-8. doi: 10.1097/00007632-199606010-00011. PMID 8725925
- [Background] Williamson E. Fear Avoidance Beliefs Questionnaire (FABQ). Aust J Physiother. 2006;52(2):149. doi: 10.1016/s0004-9514(06)70052-6. No abstract available. PMID 16805041
- [Background] Jensen LD, Maribo T, Schiottz-Christensen B, Madsen FH, Gonge B, Christensen M, Frost P. Counselling low-back-pain patients in secondary healthcare: a randomised trial addressing experienced workplace barriers and physical activity. Occup Environ Med. 2012 Jan;69(1):21-8. doi: 10.1136/oem.2010.064055. Epub 2011 May 19. PMID 21597108